CLINICAL TRIAL: NCT00390832
Title: Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of Erythropoietin in Patients With ST-Segment-Elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention (REVIVAL-3)
Brief Title: Efficacy Study of Erythropoietin After Revascularization in Myocardial Infarction (REVIVAL-3)
Acronym: REVIVAL-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Prof. A. Schömig, Deutsches Herzzentrum Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. I01106
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2009-03

CONDITIONS: Myocardial Infarction; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: STEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Erythropoietin; epoetin beta; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): recombinant human erythropoietin beta
  Interventions: Drug: Erythropoietin
- B (Placebo Comparator): 0.9% NaCl solution
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Erythropoietin — 33.333 IU of recombinant human erythropoietin beta are given at 3 time points (immediately, 24 hours and 48 hours after percutaneous coronary intervention) providing a cumulative dose of 100.000 IU
  Other Names: NeoRecormon
  Arms: A
Other: Placebo — Patients will receive placebo immediately, 24 hours and 48 hours after percutaneous coronary intervention.
  Other Names: 0.9% NaCl
  Arms: B

SUMMARY:
The purpose of this study is to determine whether erythropoietin is superior to placebo with respect to left ventricular ejection fraction in patients with ST-elevation myocardial infarction undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
Erythropoietin has lately been shown to exert others than merely hematopoietic functions. Due to attenuation of cell apoptosis and necrosis and/or enhancing neovascularisation, erythropoietin could be protective after myocardial ischemia and reperfusion and lead to infarct size reduction and improvement in left ventricular function. In a controlled clinical trial, short-term administration of erythropoietin in patients with ischemic stroke was associated with a significantly better functional recovery, with a lower level of circulating damage markers and a strong trend to smaller infarct sizes measured by magnetic resonance imaging. While leaving hematocrit and platelet counts unchanged, short-term administration of erythropoietin was shown to be safe and very well tolerated (no side effects reported or observed). The protective effects of short-term erythropoietin in acute ischemic brain damage are further evaluated in an ongoing multi-center trial in Germany. Considering the preclinical and clinical data erythropoietin is an attractive candidate to be evaluated in patients with acute myocardial infarction. In a pilot trial enrolling 22 patients with acute myocardial infarction short-term administration of erythropoietin was shown to be safe and to significantly increase the level of endothelial progenitor cells after percutaneous coronary intervention. However, the very small population did not allow evaluating the benefit in left ventricular function or clinical outcomes.

The aim of the REVIVAL-3 study is to investigate whether there is additional benefit of short-term administration of erythropoietin in patients with acute myocardial infarction after successful primary percutaneous coronary intervention (PCI) in terms of left ventricular ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-Segment elevation myocardial infarction <24 h from pain onset
* Successful primary PCI and left ventricular ejection fraction <50%
* Informed, written consent
* In women with childbearing potential a pregnancy test is mandatory

Exclusion Criteria:

* Age < 18 and > 80 years
* Cardiogenic shock
* pericarditis
* thrombolysis for the index infarction
* malignancies/other comorbid conditions with life expectancy < 1 year
* previous myocardial infarction
* planned staged PCI or prior PCI within 30 days from index procedure
* uncontrolled hypertension >160/100mmHg unresponsive to therapy
* epilepsy
* active bleeding; bleeding diathesis; history of gastrointestinal or genitourinary bleeding, recent trauma or major surgery < 1 month; history of intracranial bleeding or structural abnormalities; suspected aortic dissection; patient's refusal to blood transfusion
* hematologic disorders such as essential thrombocytosis, megakaryoblastic leukemia, polycythemia vera
* relevant hematologic deviations: hemoglobin < 100 g/l or hemoglobin > 160 g/l platelet count < 100 x 10^9 cells/l or platelet count > 600 x 10^9 cells/l
* any contraindication to magnetic resonance imaging: electronically, magnetically and mechanically activated implants such as cardiac pacemakers, automatic cardioverter defibrillators, joint prostheses, surgical/vascular clips/ hearing aids, neurostimulators, infusion pumps etc metallic splinters in the eye ferromagnetic haemostatic clips in the central nervous system cochlear implants lead wires or similar wires prosthetic heart valves, if dehiscence is suspected non-ferromagnetic stapedial implants, hemostatic clips
* glomerular filtration rate < 30 ml/min or serum creatinine > 30 mg/l or dependence on renal dialysis
* chronic liver disease with GOT > 5-fold over the normal range
* allergy to erythropoietin/true anaphylaxis after prior exposure to contrast media
* phenylketonuria
* previous enrollment in this trial
* women who are known to be pregnant, who are of childbearing potential and test positive for pregnancy, who have given birth within the last 90 days, who are breastfeeding
* patient's inability to fully cooperate with the study protocol
* other contraindication according to the summary of product characteristics of recombinant human erythropoietin beta (NeoRecormon®)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction measured by magnetic resonance imaging | 4-6 months

SECONDARY OUTCOMES:
Changes in left ventricular ejection fraction and infarct size | over 6 months
Death, recurrent myocardial infarction, IRA-revascularization and stroke | 30 days, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schomig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Ilka Ott, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - 1. Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Kastrati A, Mehilli J, Dirschinger J, Schricke U, Neverve J, Pache J, Martinoff S, Neumann FJ, Nekolla S, Blasini R, Seyfarth M, Schwaiger M, Schomig A; Stent versus Thrombolysis for Occluded Coronary Arteries in Patients With Acute Myocardial Infarction (STOPAMI-2) Study. Myocardial salvage after coronary stenting plus abciximab versus fibrinolysis plus abciximab in patients with acute myocardial infarction: a randomised trial. Lancet. 2002 Mar 16;359(9310):920-5. doi: 10.1016/S0140-6736(02)08022-4. PMID 11918909
- [Background] Zohlnhofer D, Hausleiter J, Kastrati A, Mehilli J, Goos C, Schuhlen H, Pache J, Pogatsa-Murray G, Heemann U, Dirschinger J, Schomig A. A randomized, double-blind, placebo-controlled trial on restenosis prevention by the receptor tyrosine kinase inhibitor imatinib. J Am Coll Cardiol. 2005 Dec 6;46(11):1999-2003. doi: 10.1016/j.jacc.2005.07.060. Epub 2005 Nov 4. PMID 16325031
- [Background] Pache J, Kastrati A, Mehilli J, Bollwein H, Ndrepepa G, Schuhlen H, Martinoff S, Seyfarth M, Nekolla S, Dirschinger J, Schwaiger M, Schomig A. A randomized evaluation of the effects of glucose-insulin-potassium infusion on myocardial salvage in patients with acute myocardial infarction treated with reperfusion therapy. Am Heart J. 2004 Jul;148(1):e3. doi: 10.1016/j.ahj.2004.01.019. PMID 15215812
- [Background] Sadamoto Y, Igase K, Sakanaka M, Sato K, Otsuka H, Sakaki S, Masuda S, Sasaki R. Erythropoietin prevents place navigation disability and cortical infarction in rats with permanent occlusion of the middle cerebral artery. Biochem Biophys Res Commun. 1998 Dec 9;253(1):26-32. doi: 10.1006/bbrc.1998.9748. PMID 9875214
- [Background] Ehrenreich H, Timner W, Siren AL. A novel role for an established player: anemia drug erythropoietin for the treatment of cerebral hypoxia/ischemia. Transfus Apher Sci. 2004 Aug;31(1):39-44. doi: 10.1016/j.transci.2004.05.001. PMID 15294194
- [Background] Ehrenreich H, Hasselblatt M, Dembowski C, Cepek L, Lewczuk P, Stiefel M, Rustenbeck HH, Breiter N, Jacob S, Knerlich F, Bohn M, Poser W, Ruther E, Kochen M, Gefeller O, Gleiter C, Wessel TC, De Ryck M, Itri L, Prange H, Cerami A, Brines M, Siren AL. Erythropoietin therapy for acute stroke is both safe and beneficial. Mol Med. 2002 Aug;8(8):495-505. PMID 12435860
- [Result] Ott I, Schulz S, Mehilli J, Fichtner S, Hadamitzky M, Hoppe K, Ibrahim T, Martinoff S, Massberg S, Laugwitz KL, Dirschinger J, Schwaiger M, Kastrati A, Schmig A; REVIVAL-3 Study Investigators. Erythropoietin in patients with acute ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention: a randomized, double-blind trial. Circ Cardiovasc Interv. 2010 Oct;3(5):408-13. doi: 10.1161/CIRCINTERVENTIONS.109.904425. Epub 2010 Aug 24. PMID 20736448
- [Derived] Steppich B, Groha P, Ibrahim T, Schunkert H, Laugwitz KL, Hadamitzky M, Kastrati A, Ott I; Regeneration of Vital Myocardium in ST-Segment Elevation Myocardial Infarction by Erythropoietin (REVIVAL-3) Study Investigators. Effect of Erythropoietin in patients with acute myocardial infarction: five-year results of the REVIVAL-3 trial. BMC Cardiovasc Disord. 2017 Jan 21;17(1):38. doi: 10.1186/s12872-016-0464-3. PMID 28109258